CLINICAL TRIAL: NCT03329443
Title: The Effect of Spironolactone on Acute Kidney Injury in Patients Undergoing Coronary Angiography
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alhasan Mujtaba Abdul-Wahid (Other)
Collaborators: Ministry of Health-Basra Health Directorate-Al-Sader Teaching Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Alhasan Mujtaba Abdul-Wahid, Clinical pharmacy specialist, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT00964
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Acute Kidney Injury; IHD; Contrast-induced Nephropathy
Keywords: spironolactone
MeSH Terms: conditions — Acute Kidney Injury | interventions — Spironolactone; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet
- Spironolactone (Active Comparator)
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone — each patient will receive 200 mg of spironolactone as per his/her angiography premedications
  Other Names: Active group
  Arms: Spironolactone
Drug: Placebo Oral Tablet — Each patient will receive a placebo tablet as per his/her angiography premedications
  Other Names: Control group
  Arms: placebo

SUMMARY:
an interventional study to measure the possible effects of spironolactone ( an aldosterone antagonist) on the incidence of acute kidney injury after coronary angiography

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to angiography unit
* over 18
* informed consent

Exclusion Criteria:

* acute renal failure before 7 days
* spironolactone contraindications
* hyperkalemia (S.K. >5.5 mEq/L)
* documented tumor
* actively taking NSAIDs, Ciclosporin, Cisplatin,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury by K-DIGO guidelines | 48-72 hrs
  an absolute elevation of serum creatinine of 0.5mg/dl or 25% above baseline

SECONDARY OUTCOMES:
acute kidney injury by NGAL | 6 hours
  assessment of serum NGAL at admission and after 6 hrs to detect possible AKI in selected patients

OTHER OUTCOMES:
safety outcome: serum potassium | 6 hrs
  serum potassium after 6 hrs of angio

CONTACTS AND LOCATIONS:
Overall Officials: Alhasan Mujtaba, BCPS, Principal Investigator — Baghdad University/College of Pharmacy/Department of Clinical Pharmacy; Mohammed A Taher, Ph.D., Study Chair — Baghdad University/College of Pharmacy/Department of Biochemistry; Mazin A Hazzaa', Ph.D., Study Director — Al-Sader teaching Hospital/Basra Cardiac Center/M.D. Cardiologist; Hassan M Al Rubaye, Ph.D, Study Director — Al-Sader teaching Hospital/Basra Cardiac Center/M.D. Cardiologist; Assad H Kata, Ph.D, Study Director — Al-Sader teaching Hospital/Basra Cardiac Center/M.D. Cardiologist; Hayder K Abdullkreem, M.Sc, Study Director — Head of the clinical laboratory department/ Al-Sader teaching hopital; Hamid A Abdulsada, Ph.D, Study Director — Al-Sader teaching Hospital/Basra Cardiac Center/M.D. Cardiologist; Abdul Ameer A Abdul Hameed, PH.D, Study Director — Al-Sader teaching Hospital/Basra Cardiac Center/M.D. Cardiologist
Locations (1):
- Al-Sader Teaching Hospital, Basra, Iraq

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mujtaba A, Taher MA, Hazza MA, Al-Rubaye HM, Kata AH, AbdulWahab H, AbdulBari A, AlRubay HK. The Effect of Spironolactone on the Incidence of Contrast-Induced Nephropathy in Patients Undergoing Cardiac Catheterization: Study Design and Rationale. Cardiol Ther. 2018 Jun;7(1):101-106. doi: 10.1007/s40119-018-0112-3. Epub 2018 May 21. PMID 29785539